CLINICAL TRIAL: NCT01724437
Title: Unexcitability Along the Ablation as an Endpoint for Atrial Fibrillation Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PV3503
Record Dates: First submitted 2012-11-04; First posted 2012-11-09 (Estimated); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Paroxysmal Atrial Fibrillation; Catheter Ablation Strategies
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Masking Description: Open Label

ARMS (2):
- Loss of pace capture (Active Comparator): Pulmonary vein isolation: Ablation along the ablation line is continued until loss of pace capture along the ablation line is achieved
  catheter based pulmonary vein isolation
  Interventions: Device: catheter based pulmonary vein isolation
- Conventional (Active Comparator): Pulmonary vein isolation: Ablation is discontinued when electrical isolation of the pulmonary veins is achieved.
  catheter based pulmonary vein isolation
  Interventions: Device: catheter based pulmonary vein isolation

INTERVENTIONS:
Device: catheter based pulmonary vein isolation — catheter based ablation using irrigated catheters and radiofrequency energy as in clinical practice

SUMMARY:
to assess the near-term (12 months) efficacy of pulmonary vein isolation.

DETAILED DESCRIPTION:
The aim of the study was to assess the near-term (12 months) efficacy of pulmonary vein isolation using a standard approach compared to application of an additional acute procedural endpoint of unexcitability along the ablation line.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* age > 18 years
* paroxysmal atrial fibrillation

Exclusion Criteria:

* structural heart disease
* intracardiac thrombus
* reversible causes of atrial fibrillation
* inability to take warfarin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
time to AF and AT recurrence | 12 months
  recurrence of AF as assessed by 3 day holter monitoring, assessment of AT recurrence using 3 day holter monitoring

SECONDARY OUTCOMES:
procedure duration | completed (15 months)
  time needed to complete the procedure
procedure safety | up to three days after the procedure
  complication such as groin hematoma, stroke and pericardial bleed prolonging the hospital stay will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Willems, Principal Investigator — Universitäres Herzzentrum Hamburg GmbH
Locations (1):
- University Hospital Hamburg, Hamburg, Germany

REFERENCES:
- [Derived] Steven D, Sultan A, Reddy V, Luker J, Altenburg M, Hoffmann B, Rostock T, Servatius H, Stevenson WG, Willems S, Michaud GF. Benefit of pulmonary vein isolation guided by loss of pace capture on the ablation line: results from a prospective 2-center randomized trial. J Am Coll Cardiol. 2013 Jul 2;62(1):44-50. doi: 10.1016/j.jacc.2013.03.059. Epub 2013 May 1. PMID 23644091